CLINICAL TRIAL: NCT00074152
Title: A Randomized Clinical Trial Of Adjuvant Chemotherapy For Radically Resected Loco-Regional Relapse Of Breast Cancer
Brief Title: Adjuvant Chemotherapy in Treating Women Who Have Undergone Resection for Relapsed Breast Cancer; Chemotherapy as Adjuvant for LOcally Recurrent Breast Cancer
Acronym: CALOR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ETOP IBCSG Partners Foundation (Network)
Collaborators: NSABP Foundation Inc (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000343619; IBCSG-27-02 (Other: IBCSG); BIG-1-02 (Other: Breast International Group); EU-20320; NSABP-B-37; 2005-001484-64 (EudraCT Number)
Record Dates: First submitted 2003-12-10; First posted 2003-12-11 (Estimated); Results first posted 2015-05-12 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-05

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Drug Therapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Active Comparator): Patients receive radiotherapy* within 6 months after surgery.
  Interventions: Radiation: radiation therapy
- Arm II (Experimental): Within 10 weeks after surgery, patients receive at least 3 courses of an adjuvant chemotherapy regimen as determined by the investigator. Patients may receive radiotherapy within 6 months after surgery and after the completion of chemotherapy OR integrated with chemotherapy.
  Interventions: Drug: chemotherapy

INTERVENTIONS:
Drug: chemotherapy — Given within 10 weeks after surgery.
  Arms: Arm II
Radiation: radiation therapy — Given within 6 months after surgery
  Arms: Arm I

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known whether chemotherapy is effective in treating women who have undergone surgery and radiation therapy for relapsed breast cancer.

PURPOSE: Randomized phase III trial to determine the effectiveness of adjuvant chemotherapy in treating women who have undergone resection for local and/or regional relapsed breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of adjuvant chemotherapy, in terms of disease-free survival, in women with radically resected loco-regional relapsed breast cancer.

Secondary

* Determine the systemic disease-free and overall survival of patients treated with this regimen.
* Determine the sites of recurrence, incidence of second (non-breast) malignancies, and causes of death without relapse of breast cancer in patients treated with this regimen.
* Determine the quality of life of patients treated with this regimen (QOL portion closed 11/13/08).

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to prior chemotherapy (yes vs no), estrogen receptor (ER) positive and/or progesterone receptor (PR) positive (yes vs no), and location of recurrence (breast vs mastectomy scar/chest wall vs regional lymph nodes). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive radiotherapy* within 6 months after surgery.
* Arm II: Within 10 weeks after surgery, patients receive at least 3 courses of an adjuvant chemotherapy regimen as determined by the investigator. Patients also receive radiotherapy* within 6 months after surgery and after the completion of chemotherapy OR integrated with chemotherapy.

NOTE: *Patients with clear margins (R0) who received prior adjuvant radiotherapy are not required to receive further radiotherapy

Patients with ER and/or PR positive tumors also receive standard hormonal therapy.

Quality of life is assessed at baseline and at 9 and 12 months (QOL portion closed 11/13/08).

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 265 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive breast cancer

  * First local and/or regional (i.e., ipsilateral axillary or internal mammary lymph node region) recurrence after primary treatment with mastectomy or lumpectomy/quadrantectomy with clear surgical margins

    * Local failure is defined as a tumor recurrence in any soft tissue of the ipsilateral conserved breast or the chest wall, mastectomy scar, and/or skin
    * Regional failure is defined as a tumor recurrence in the ipsilateral axillary lymph nodes, extranodal soft tissue of the ipsilateral axilla, and/or ipsilateral internal mammary. Regional failure does not include supraclavicular lymph nodes or tumor in the opposite breast
  * No other prior recurrence in any site, including local
* Surgical resection of the recurrence meeting 1 of the following criteria:

  * Uninvolved ("clear") margins and planned radiotherapy with at least 40 Gy for patients who had no prior adjuvant radiotherapy
  * Mastectomy of the recurrence with uninvolved ("clear") margins after lumpectomy/quadrantectomy alone for the primary
* Adjuvant trastuzumab (Herceptin®) therapy or other HER-2 directed therapies are allowed for patients with HER-2 positive tumors and must be declared prior to randomization
* No evidence of distant metastasis, including ipsilateral supraclavicular lymph nodes, by x-ray or CT scan of the chest, ultrasound or CT scan of the abdomen and pelvis, or bone scintigraphy only if alkaline phosphatase is > 2 times normal or if medically indicated (e.g., bone pain)
* No macroscopically incomplete surgery
* No bilateral malignancy except carcinoma in situ
* No suspicious mass in the opposite breast unless that mass has been proven by biopsy to be benign
* No skeletal pain of unknown cause

  * No hot spots on bone scan for which metastases cannot be ruled out by x-ray, MRI, and/or CT scan
* Hormone receptor status:

  * Determined in the recurrent tumor by immunohistochemistry and/or ligand-binding assay
  * Estrogen receptor positive or negative
  * Progesterone receptor positive or negative

PATIENT CHARACTERISTICS:

Age

* Minimum 18 years

Sex

* Female

Menopausal status

* Not specified

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* No elevated alkaline phosphatase

Renal

* Not specified

Other

* Fertile patients must use effective non-hormonal contraception
* Medically suitable for chemotherapy of 3-6 months duration
* No other primary malignant tumors except adequately treated carcinoma in situ of the cervix or nonmelanoma skin cancer
* No non-malignant systemic disease that would preclude study treatment or prolong follow-up
* No psychiatric or addictive disorder that would preclude giving informed consent
* No history of noncompliance to medical regimens or potential for being unreliable

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics

Surgery

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2002-07; Primary Completion 2014-02 (Actual); Study Completion 2016-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Aebi, MD, Study Chair — Inselspital Bern, Switzerland; Irene L. Wapnir, MD, Study Chair — Stanford Cancer Center, CA, USA
Locations (199):
- United States (166):
  - Kaiser Permanente - Deer Valley, Antioch, California
  - Kaiser Permanente - Fremont, Fremont, California
  - Kaiser Permanente Medical Center - Hayward, Hayward, California
  - Kaiser Permanente Medical Center - Oakland, Oakland, California
  - Kaiser Permanente Medical Center - Redwood City, Redwood City, California
  - Kaiser Permanente Medical Center - Richmond, Richmond, California
  - Kaiser Permanente Medical Center - Roseville, Roseville, California
  - South Sacramento Kaiser-Permanente Medical Center, Sacramento, California
  - Kaiser Permanente Medical Center - Sacramento, Sacramento, California
  - Kaiser Permanente Medical Center - San Francisco Geary Campus, San Francisco, California
  - Kaiser Permanente Medical Center - Santa Teresa, San Jose, California
  - Kaiser Foundation Hospital - San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara Kiely Campus, Santa Clara, California
  - Kaiser Permanente Medical Center - Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Medical Center - South San Francisco, South San Francisco, California
  - Stanford Cancer Center, Stanford, California
  - Kaiser Permanente Medical Facility - Stockton, Stockton, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California
  - Kaiser Permanente Medical Center - Walnut Creek, Walnut Creek, California
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Kent General Hospital, Dover, Delaware
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - La Grange Memorial Hospital, La Grange, Illinois
  - Edward Hospital Cancer Center, Naperville, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - Genesis Medical Center - West Campus, Davenport, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - Tufts-NEMC Cancer Center, Boston, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - Hope A Women's Cancer Center, Asheville, North Carolina
  - Batte Cancer Center at Northeast Medical Center, Concord, North Carolina
  - Southeastern Medical Oncology Center - Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Wood County Oncology Center, Bowling Green, Ohio
  - Aultman Cancer Center at Aultman Hospital, Canton, Ohio
  - MetroHealth Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - North Coast Cancer Care - Clyde, Clyde, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Kaiser Permanente Health Care - Portland, Portland, Oregon
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Western Pennsylvania Cancer Institute at Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - Hematology and Oncology Associates of Northeastern Pennsylvania, Scranton, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - AnMed Cancer Center, Anderson, South Carolina
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Christine LaGuardia Phillips Cancer Center at Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - Doctor's Hospital of Laredo, Laredo, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Danville Regional Medical Center, Danville, Virginia
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Southwest Virginia Regional Cancer Center at Wellmonth Health, Norton, Virginia
  - Community Comprehensive Cancer Center at Camden-Clark Memorial Hospital, Parkersburg, West Virginia
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - Marshfield Clinic at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Saint Michael's Hospital Cancer Center, Stevens Point, Wisconsin
  - Marshfield Clinic - Wausau Center, Wausau, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming
- Australia (5):
  - Mater Hospital - North Sydney, North Sydney, New South Wales
  - Flinders Medical Centre, Bedford Park, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria
  - Maroondah Hospital, East Ringwood, Victoria
- Institut Jules Bordet, Brussels, Belgium
- Canada (8):
  - Tom Baker Cancer Centre - Calgary, Calgary, Alberta
  - Cross Cancer Institute at University of Alberta, Edmonton, Alberta
  - Edmond Odette Cancer Centre at Sunnybrook, Toronto, Ontario
  - Hopital Notre-Dame du CHUM, Montreal, Quebec
  - CHUM - Hotel Dieu Hospital, Montreal, Quebec
  - CHUM - Hopital Saint-Luc, Montreal, Quebec
  - Jewish General Hospital - Montreal, Montreal, Quebec
  - Hopital du Saint-Sacrement - Quebec, Québec, Quebec
- National Institute of Oncology, Budapest, Hungary
- Netherlands (4):
  - Arnhems Radiotherapeutisch Instituut, Arnhem
  - Leiden University Medical Center, Leiden
  - Universitair Medisch Centrum St. Radboud - Nijmegen, Nijmegen
  - Isala Klinieken - locatie Sophia, Zwolle
- Instituto Nacional de Enfermedades Neoplasicas, Lima, Peru
- Groote Schuur Hospital, Cape Town, South Africa
- Spain (7):
  - Hospital Universitario Puerta Del Mar, Cadiz
  - Hospital Cuidad de Jaen, Jaén
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitario San Carlos, Madrid
  - Fundacion Hospital Alcorcon, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Clinico Universitario de Valencia, Valencia
- Switzerland (5):
  - Inselspital Bern, Bern
  - Ospedale Beata Vergine, Mendrisio
  - Kantonsspital - St. Gallen, Sankt Gallen
  - Regionalspital, Thun
  - Klinik und Poliklinik fur Gynakologie, Zurich, Zurich

REFERENCES:
- [Result] Wapnir IL, Aebi S, Gelber S, Anderson SJ, Lang I, Robidoux A, Mamounas EP, Wolmark N. Progress on BIG 1-02/IBCSG 27-02/NSABP B-37, a prospective randomized trial evaluating chemotherapy after local therapy for isolated locoregional recurrences of breast cancer. Ann Surg Oncol. 2008 Nov;15(11):3227-31. doi: 10.1245/s10434-008-0129-2. Epub 2008 Sep 11. PMID 18784962
- [Result] Wapnir IL, Aebi S, Geyer CE, Zahrieh D, Gelber RD, Anderson SJ, Robidoux A, Bernhard J, Maibach R, Castiglione-Gertsch M, Coates AS, Piccart MJ, Clemons MJ, Costantino JP, Wolmark N; IBCSG; BIG; NSABP. A randomized clinical trial of adjuvant chemotherapy for radically resected locoregional relapse of breast cancer: IBCSG 27-02, BIG 1-02, and NSABP B-37. Clin Breast Cancer. 2008 Jun;8(3):287-92. doi: 10.3816/CBC.2008.n.035. PMID 18650162
- [Result] Aebi S, Gelber S, Anderson SJ, Lang I, Robidoux A, Martin M, Nortier JW, Paterson AH, Rimawi MF, Canada JM, Thurlimann B, Murray E, Mamounas EP, Geyer CE Jr, Price KN, Coates AS, Gelber RD, Rastogi P, Wolmark N, Wapnir IL; CALOR investigators. Chemotherapy for isolated locoregional recurrence of breast cancer (CALOR): a randomised trial. Lancet Oncol. 2014 Feb;15(2):156-63. doi: 10.1016/S1470-2045(13)70589-8. Epub 2014 Jan 16. PMID 24439313
- [Derived] Wapnir IL, Price KN, Anderson SJ, Robidoux A, Martin M, Nortier JWR, Paterson AHG, Rimawi MF, Lang I, Baena-Canada JM, Thurlimann B, Mamounas EP, Geyer CE Jr, Gelber S, Coates AS, Gelber RD, Rastogi P, Regan MM, Wolmark N, Aebi S; International Breast Cancer Study Group; NRG Oncology, GEICAM Spanish Breast Cancer Group, BOOG Dutch Breast Cancer Trialists' Group; Breast International Group. Efficacy of Chemotherapy for ER-Negative and ER-Positive Isolated Locoregional Recurrence of Breast Cancer: Final Analysis of the CALOR Trial. J Clin Oncol. 2018 Apr 10;36(11):1073-1079. doi: 10.1200/JCO.2017.76.5719. Epub 2018 Feb 14. PMID 29443653

RESULTS

PARTICIPANT FLOW:
Groups:
- Observation: Observation (+/- Radiation). Patients receive radiotherapy* within 6 months after surgery.
  radiation therapy: Given within 6 months after surgery
- Chemotherapy: Chemotherapy (+/- Radiation). Within 10 weeks after surgery, patients receive at least 3 courses of an adjuvant chemotherapy regimen as determined by the investigator. Patients may receive radiotherapy within 6 months after surgery and after the completion of chemotherapy OR integrated with chemotherapy.
  chemotherapy: Given within 10 weeks after surgery.
Period: Overall Study
Arm/Group | Observation | Chemotherapy
Started | 77 | 85
Completed | 22 | 52
Not Completed | 55 | 33
Not completed — Death | 21 | 9
Not completed — Lack of Efficacy | 34 | 24

BASELINE CHARACTERISTICS:
Groups:
- Arm I: Observation (+/- Radiation). Patients receive radiotherapy* within 6 months after surgery.
  radiation therapy: Given within 6 months after surgery
- Arm II: Chemotherapy (+/- Radiation). Within 10 weeks after surgery, patients receive at least 3 courses of an adjuvant chemotherapy regimen as determined by the investigator. Patients may receive radiotherapy within 6 months after surgery and after the completion of chemotherapy OR integrated with chemotherapy.
  chemotherapy: Given within 10 weeks after surgery.
- Total: Total of all reporting groups
Arm/Group | Arm I | Arm II | Total
Number analyzed (Participants) | 77 | 85 | 162
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 60 | 71 | 131
  >=65 years | 17 | 14 | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 85 | 162
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 23 | 42
  Hungary | 17 | 16 | 33
  Canada | 15 | 16 | 31
  Spain | 9 | 11 | 20
  Peru | 1 | 0 | 1
  Australia | 1 | 1 | 2
  South Africa | 3 | 2 | 5
  Netherlands | 6 | 6 | 12
  Switzerland | 6 | 10 | 16
Prior chemotherapy [Number; unit: participants]
  Yes | 52 | 49 | 101
  No | 25 | 36 | 61
Surgery for primary tumor [Number; unit: participants]
  Mastectomy | 31 | 33 | 64
  Breast conserving | 46 | 52 | 98
Estrogen receptor (ER) status of the isolated local or regional recurrence [Number; unit: participants]
  Positive | 48 | 56 | 104
  Negative | 29 | 29 | 58
Progesterone receptor (PgR) status of the isolated local or regional recurrence [Number; unit: participants]
  positive | 35 | 44 | 79
  negative | 40 | 39 | 79
  not available | 2 | 2 | 4
Location of isolated loco-regional recurrence (ILRR) [Number; unit: participants]
  Breast | 41 | 47 | 88
  Mx scar/chest wall | 26 | 27 | 53
  Regional lymph nodes | 10 | 11 | 21
Menopausal Status at isolated loco-regional recurrence (ILRR) [Number; unit: participants]
  pre | 14 | 20 | 34
  post | 63 | 65 | 128
Time from primary surgery to isolated loco-regional recurrence (ILRR) surgery [Median (Full Range); unit: years] | 6.2 [2.9 to 11.3] | 5.0 [2.9 to 9.5] | 5.5 [2.9 to 11.3]
Estrogen receptor (ER) status of primary tumor [Number; unit: participants]
  negative | 20 | 27 | 47
  positive | 47 | 49 | 96
  unknown | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival
Time Frame: 5 years after randomization
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 77 | 85
percentage of participants | 57 [44 to 67] | 69 [56 to 79]

2. Secondary Outcome: Overall Survival
Time Frame: 5 years after randomization
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Arm I: Observation (+/- Radiation).Patients receive radiotherapy* within 6 months after surgery.
  radiation therapy: Given within 6 months after surgery
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 77 | 85
percentage of participants | 76 [63 to 85] | 88 [77 to 94]

3. Secondary Outcome: Sites of First Failures
Description: Tumor recurrence in the breast, lymph nodes or other areas of the body including bone, lung, liver, central nervous system, bone marrow
Time Frame: 5 years after randomization
Measure: Number; unit: participants
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 77 | 85
participants
  Failures | 34 | 24
  Deaths | 21 | 9
  Local or Regional | 9 | 6
  Distant | 22 | 15
  Soft Tissue | 2 | 0
  Bone | 5 | 8
  Viscera | 15 | 7
  Contralateral Breast | 1 | 1
  Secon (non-breast) Malignancy | 0 | 1
  Death without prior Cancer Event | 0 | 1
  Death, cause unknown | 2 | 0

ADVERSE EVENTS:
Time Frame: From date patient provided informed consent until 4 weeks after study treatment completion, beyond 4 weeks after stopping study treatment any death or serious adverse event considered possibly related to previous study treatment (approximately 10 years)
Arm/Group | Arm I | Arm II
Serious Adverse Events (participants affected / at risk) | 0/77 | 12/85
Other Adverse Events (participants affected / at risk) | 0/77 | 0/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=77) | Arm II (N=85)
Febrile neutropenia (Infections and infestations) | 0 (0) | 3 (3)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Pulmonary/upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Neutropenia with symptoms of generalized musculoskeletal pain and fatigue
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cardiac ischemia (Cardiac disorders) | 0 (0) | 2 (2)
Motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Endometrial mucosa thinkening (Reproductive system and breast disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No